CLINICAL TRIAL: NCT02346435
Title: The Delayed Intervention and Surveillance for Small Renal Masses (DISSRM) Registry
Acronym: DISSRM
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Other Study IDs: 17821; NA_00016036 (Other: AbramsonCC); 850179 (Other: UPenn IRB)
Record Dates: First submitted 2014-06-06; First posted 2015-01-27 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Kidney Neoplasm
Keywords: small renal mass; active surveillance
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Active Surveillance
- Immediate Intervention: May include patients undergoing open or minimally-invasive partial nephrectomy, radical nephrectomy or energy ablation.
- Crossover (Delayed Intervention): Initially patients in active surveillance that meet progression criteria or elect to undergo delayed intervention.

SUMMARY:
Retrospective studies indicate that active surveillance for clinically localized, small renal masses (cT1a, <=4cm) is safe. It is our hypothesis that active surveillance is safe and efficacious when compared prospectively to patients undergoing immediate intervention for their small renal mass.

DETAILED DESCRIPTION:
All patients are offered active surveillance or immediate intervention, as applicable, prior to being offered consent for the DISSRM Registry. All patients are enrolled and followed prospectively. Surveillance patients are followed per protocol with serial imaging, blood work and quality of life questionnaires. Intervention patients are followed at the discretion of the attending surgeon with serial QOL appointments/questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must have a solid, enhancing renal mass ≤4cm at its greatest dimension found on incidental scanning in the last 6 months.
* Age ≥ 18 and able to read, understand and sign informed consent.
* Must be willing to adhere to the treatment algorithm and time constraints therein.

Exclusion Criteria:

* Cannot have suspicion of metastases to the kidney if any other malignancy diagnosed within two years of study entry.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients (18-100) presenting with a clinically localized, solid renal mass (cT1a, <=4cm).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Disease-specific survival | 5 years
  Safety and Efficacy of active surveillance and delayed intervention for the SRM, measured by disease-free survival at 5-years.

SECONDARY OUTCOMES:
Objective Safety and Tolerability of Percutaneous Renal Biopsy | 5 years
  Measured by observed total (minor and major) complications compared to historical complication rates for this procedure.
Quality-of-life outcomes for patients undergoing AS versus definitive therapy. | 5 years
  Measured by SF12 Questionnaire at enrollment, 6 and 12 months and annually thereafter.
To determine objective selection criteria for active surveillance. | 5 years
  Demographic (i.e. age, sex, race), clinical (i.e. comorbidities, medications, family history) and imaging characteristics (i.e. tumor size, enhancement patterns, tumor complexity) will be used to determine patients most suitable for active surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Allaf, MD, MBA, Principal Investigator — Johns Hopkins University; Nirmish Singla, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States